CLINICAL TRIAL: NCT00766584
Title: Autonomic Nervous System Activity, Aging and Sleep Apnea/Hypopnea in a Prospective Cohort of Subjects Aged 67 Years
Brief Title: Autonomic Nervous System Activity, Aging and Sleep Apnea/Hypopnea
Acronym: SYNAPSE
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0201085; DGS 2003/0069
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Aging; Autonomic nervous system; stroke; Myocardiac infarction; Prospective cohort; Sleep apnea/hypopnea
MeSH Terms: conditions — Stroke; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROOF cohort: This cohort is the same than the PROOF study (NCT00759304). Subjects were recruited amongst the inhabitants of the city of Saint-Etienne, France, and were eligible if aged 65 at the inclusion date in the PROOF study
  Interventions: Other: Sleep apnea/hypopnea detection

INTERVENTIONS:
Other: Sleep apnea/hypopnea detection — Simultaneous 24-hour ambulatory electrocardiogram and polygraphic recordings performed at home during a night.
  Other Names: HypnoPTT, Tyco Healthcare, USA

SUMMARY:
The regulatory effects of the autonomic nervous system (ANS) concern almost all organs which permanently feed information back to this global biological vigilance system controlling allostasis. Heart rate fluctuations are highly dependent on ANS control, making the heart one of the best indicators of ANS activity.

Low ANS activity level is associated with severe cardiac and cerebral events, as well as to death from any cause in the general population. It is even associated with sleep apnea/hypopnea.

DETAILED DESCRIPTION:
The main goal of this SYNAPSE study is to evaluate, on a selected prospective cohort of subjects aged 67 years upon study entry, the incidence of sleep apnea/hypopnea and the prognostic values of ANS activity levels measured at preset times and of cardiovascular or cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* to participate in the PROOF study

Exclusion Criteria:

* prior myocardiac infarction
* prior stroke
* hearth failure
* atrial fibrillation
* insulin-treated diabetes mellitus
* cardiac pacemaker
* disease limiting life expectancy to < 5 years
* contraindication to brain MRI
* living in an institution
* respiratory failure with oxygenotherapy
* sleep-related breathing disorders known and treated

Ages: 67 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects were recruited amongst the inhabitants of the city of Saint-Etienne, France, and were eligible if aged 65 at the inclusion date in the PROOF study
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2003-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite criterion : fatal and non-fatal cardiovascular or cerebrovascular events | During all the study

SECONDARY OUTCOMES:
Presence and relationship of sleep apnea/hypopnea and clinically silent stroke revealed through brain MRI | Years 1, 3, 5, 7 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARTHELEMY, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsuji H, Venditti FJ Jr, Manders ES, Evans JC, Larson MG, Feldman CL, Levy D. Reduced heart rate variability and mortality risk in an elderly cohort. The Framingham Heart Study. Circulation. 1994 Aug;90(2):878-83. doi: 10.1161/01.cir.90.2.878. PMID 8044959
- [Background] Pitson DJ, Stradling JR. Autonomic markers of arousal during sleep in patients undergoing investigation for obstructive sleep apnoea, their relationship to EEG arousals, respiratory events and subjective sleepiness. J Sleep Res. 1998 Mar;7(1):53-9. doi: 10.1046/j.1365-2869.1998.00092.x. PMID 9613428
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Lavie P, Lavie L, Herer P. All-cause mortality in males with sleep apnoea syndrome: declining mortality rates with age. Eur Respir J. 2005 Mar;25(3):514-20. doi: 10.1183/09031936.05.00051504. PMID 15738297
- [Result] Barthelemy JC, Pichot V, Dauphinot V, Celle S, Laurent B, Garcin A, Maudoux D, Kerleroux J, Lacour JR, Kossovsky M, Gaspoz JM, Roche F. Autonomic nervous system activity and decline as prognostic indicators of cardiovascular and cerebrovascular events: the 'PROOF' Study. Study design and population sample. Associations with sleep-related breathing disorders: the 'SYNAPSE' Study. Neuroepidemiology. 2007;29(1-2):18-28. doi: 10.1159/000108914. PMID 17898520
- [Result] Celle S, Peyron R, Faillenot I, Pichot V, Alabdullah M, Gaspoz JM, Laurent B, Barthelemy JC, Roche F. Undiagnosed sleep-related breathing disorders are associated with focal brainstem atrophy in the elderly. Hum Brain Mapp. 2009 Jul;30(7):2090-7. doi: 10.1002/hbm.20650. PMID 18781591
- [Derived] Sforza E, Millasseau S, Hupin D, Barthelemy JC, Roche F. Arterial stiffness alteration and obstructive sleep apnea in an elderly cohort free of cardiovascular event history: the PROOF cohort study. Sleep Breath. 2019 Mar;23(1):201-208. doi: 10.1007/s11325-018-1683-x. Epub 2018 Jun 26. PMID 29946946
- [Derived] Monneret D, Barthelemy JC, Hupin D, Maudoux D, Celle S, Sforza E, Roche F. Serum lipid profile, sleep-disordered breathing and blood pressure in the elderly: a 10-year follow-up of the PROOF-SYNAPSE cohort. Sleep Med. 2017 Nov;39:14-22. doi: 10.1016/j.sleep.2017.07.028. Epub 2017 Sep 18. PMID 29157582
- [Derived] Saint Martin M, Labeix P, Garet M, Thomas T, Barthelemy JC, Collet P, Roche F, Sforza E. Does Subjective Sleep Affect Bone Mineral Density in Older People with Minimal Health Disorders? The PROOF Cohort. J Clin Sleep Med. 2016 Nov 15;12(11):1461-1469. doi: 10.5664/jcsm.6266. PMID 27655463
- [Derived] Sforza E, Saint Martin M, Thomas T, Collet P, Garet M, Barthelemy JC, Roche F. Risk factors of osteoporosis in healthy elderly with unrecognized obstructive sleep apnea: role of physical activity. Sleep Med. 2016 Jun;22:25-32. doi: 10.1016/j.sleep.2016.04.010. Epub 2016 Jun 7. PMID 27544832
- [Derived] Sforza E, Saint Martin M, Barthelemy JC, Roche F. Mood disorders in healthy elderly with obstructive sleep apnea: a gender effect. Sleep Med. 2016 Mar;19:57-62. doi: 10.1016/j.sleep.2015.11.007. Epub 2015 Nov 25. PMID 27198948
- [Derived] Boutet C, Vassal F, Celle S, Schneider FC, Barthelemy JC, Laurent B, Barral FG, Roche F. Incidental findings on brain magnetic resonance imaging in the elderly:the PROOF study. Brain Imaging Behav. 2017 Feb;11(1):293-299. doi: 10.1007/s11682-016-9519-4. PMID 26843003
- [Derived] Sforza E, Celle S, Saint-Martin M, Barthelemy JC, Roche F. Hippocampus volume and subjective sleepiness in older people with sleep-disordered breathing: a preliminary report. J Sleep Res. 2016 Apr;25(2):190-3. doi: 10.1111/jsr.12367. Epub 2015 Dec 14. PMID 26662175
- [Derived] Sforza E, Pichot V, Martin MS, Barthelemy JC, Roche F. Prevalence and determinants of subjective sleepiness in healthy elderly with unrecognized obstructive sleep apnea. Sleep Med. 2015 Aug;16(8):981-6. doi: 10.1016/j.sleep.2015.03.010. Epub 2015 Apr 15. PMID 26141008
- [Derived] Sforza E, Sabri M, DaCosta A, Isaaz K, Barthelemy JC, Roche F. Echocardiographic Findings in Healthy Elderly People with Unrecognized Sleep Disordered Breathing. J Clin Sleep Med. 2015 Sep 15;11(9):975-80. doi: 10.5664/jcsm.5006. PMID 25902826
- [Derived] Saint Martin M, Roche F, Thomas-Anterion C, Barthelemy JC, Sforza E; PROgnostic OF cardiovascular and cerebrovascular events study group. Eight-year parallel change in baroreflex sensitivity and memory function in a sample of healthy older adults. J Am Geriatr Soc. 2015 Feb;63(2):270-5. doi: 10.1111/jgs.13252. Epub 2015 Feb 2. PMID 25641086
- [Derived] Martin MS, Sforza E, Roche F, Barthelemy JC, Thomas-Anterion C; PROOF study group. Sleep breathing disorders and cognitive function in the elderly: an 8-year follow-up study. the proof-synapse cohort. Sleep. 2015 Feb 1;38(2):179-87. doi: 10.5665/sleep.4392. PMID 25325480
- [Derived] Sforza E, Saint Martin M, Barthelemy JC, Roche F. Association of self-reported sleep and hypertension in non-insomniac elderly subjects. J Clin Sleep Med. 2014 Sep 15;10(9):965-71. doi: 10.5664/jcsm.4026. PMID 25142770
- [Derived] Saint Martin M, Sforza E, Thomas-Anterion C, Barthelemy JC, Roche F; PROOF Study Group. Baroreflex sensitivity, vascular risk factors, and cognitive function in a healthy elderly population: the PROOF cohort. J Am Geriatr Soc. 2013 Dec;61(12):2096-2102. doi: 10.1111/jgs.12548. Epub 2013 Nov 26. PMID 24279643
- [Derived] Sforza E, Thomas T, Barthelemy JC, Collet P, Roche F. Obstructive sleep apnea is associated with preserved bone mineral density in healthy elderly subjects. Sleep. 2013 Oct 1;36(10):1509-15. doi: 10.5665/sleep.3046. PMID 24082310
- [Derived] Martin MS, Sforza E, Barthelemy JC, Thomas-Anterion C, Roche F. Sleep perception in non-insomniac healthy elderly: a 3-year longitudinal study. Rejuvenation Res. 2014 Feb;17(1):11-8. doi: 10.1089/rej.2013.1457. PMID 24033249
- [Derived] Chouchou F, Pichot V, Pepin JL, Tamisier R, Celle S, Maudoux D, Garcin A, Levy P, Barthelemy JC, Roche F; PROOF Study Group. Sympathetic overactivity due to sleep fragmentation is associated with elevated diurnal systolic blood pressure in healthy elderly subjects: the PROOF-SYNAPSE study. Eur Heart J. 2013 Jul;34(28):2122-31, 2131a. doi: 10.1093/eurheartj/eht208. Epub 2013 Jun 11. PMID 23756334
- [Derived] Degache F, Sforza E, Dauphinot V, Celle S, Garcin A, Collet P, Pichot V, Barthelemy JC, Roche F; PROOF Study Group. Relation of central fat mass to obstructive sleep apnea in the elderly. Sleep. 2013 Apr 1;36(4):501-7. doi: 10.5665/sleep.2532. PMID 23564997
- [Derived] Sforza E, Gauthier M, Crawford-Achour E, Pichot V, Maudoux D, Barthelemy JC, Roche F. A 3-year longitudinal study of sleep disordered breathing in the elderly. Eur Respir J. 2012 Sep;40(3):665-72. doi: 10.1183/09031936.00133011. Epub 2012 Mar 9. PMID 22408210
- [Derived] Tonnesen P, Lauri H, Perfekt R, Mann K, Batra A. Efficacy of a nicotine mouth spray in smoking cessation: a randomised, double-blind trial. Eur Respir J. 2012 Sep;40(3):548-54. doi: 10.1183/09031936.00155811. Epub 2012 Feb 9. PMID 22323576
- [Derived] Sforza E, Chouchou F, Pichot V, Barthelemy JC, Roche F. Heart rate increment in the diagnosis of obstructive sleep apnoea in an older population. Sleep Med. 2012 Jan;13(1):21-8. doi: 10.1016/j.sleep.2011.04.011. Epub 2011 Nov 21. PMID 22104544
- [Derived] Chouchou F, Sforza E, Celle S, Pichot V, Maudoux D, Garcin A, Barthelemy JC, Roche F; PROOF Study Group. Pulse transit time in screening sleep disordered breathing in an elderly population: the PROOF-SYNAPSE study. Sleep. 2011 Aug 1;34(8):1051-9. doi: 10.5665/SLEEP.1160. PMID 21804667
- [Derived] Sforza E, Chouchou F, Collet P, Pichot V, Barthelemy JC, Roche F. Sex differences in obstructive sleep apnoea in an elderly French population. Eur Respir J. 2011 May;37(5):1137-43. doi: 10.1183/09031936.00043210. Epub 2010 Sep 3. PMID 20817711
- [Derived] Sforza E, Roche F, Thomas-Anterion C, Kerleroux J, Beauchet O, Celle S, Maudoux D, Pichot V, Laurent B, Barthelemy JC. Cognitive function and sleep related breathing disorders in a healthy elderly population: the SYNAPSE study. Sleep. 2010 Apr;33(4):515-21. doi: 10.1093/sleep/33.4.515. PMID 20394321
- [Derived] Guillot M, Costes F, Sforza E, Maudoux D, Bertoletti L, Barthelemy JC, Roche F. Is tidal expiratory flow limitation predictive of sleep-related disorders in the elderly? Eur Respir J. 2010 Oct;36(4):842-8. doi: 10.1183/09031936.00078009. Epub 2010 Apr 8. PMID 20378600